CLINICAL TRIAL: NCT00092820
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of MK0653 When Added to Current Regimen in Patients With Homozygous Sitosterolemia
Brief Title: Sitosterolemia Extension Study (0653-004)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P02243; 2004_033
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Lipid Metabolism, Inborn Errors; Heart Disease
Keywords: Homozygous Sitosterolemia
MeSH Terms: conditions — Lipid Metabolism, Inborn Errors; Heart Diseases | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653, ezetimibe
Drug: Comparator: placebo

SUMMARY:
This is an extension study for patients having unusually high absorption of non-cholesterol sterols, resulting in heart-related diseases. This study will evaluate the long term safety and the ability to lower cholesterol levels with an investigational drug.

DETAILED DESCRIPTION:
The duration of treatment is 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with elevated sitosterol levels while taking current medication

Exclusion Criteria:

* Patient has a condition which, in the opinion of the investigator, might pose a risk to the patient, interfere with participation in the study, or does not meet the additional criteria as required by the study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2001-02-12 (Actual); Primary Completion 2001-09-18 (Actual); Study Completion 2004-11-30 (Actual)

PRIMARY OUTCOMES:
Plasma sitosterol levels after 52 weeks.

SECONDARY OUTCOMES:
Plasma LDL-C and plasma campesterol. Safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Salen G, von Bergmann K, Lutjohann D, Kwiterovich P, Kane J, Patel SB, Musliner T, Stein P, Musser B; Multicenter Sitosterolemia Study Group. Ezetimibe effectively reduces plasma plant sterols in patients with sitosterolemia. Circulation. 2004 Mar 2;109(8):966-71. doi: 10.1161/01.CIR.0000116766.31036.03. Epub 2004 Feb 9. PMID 14769702
- [Background] Lutjohann D, von Bergmann K, Sirah W, Macdonell G, Johnson-Levonas AO, Shah A, Lin J, Sapre A, Musliner T. Long-term efficacy and safety of ezetimibe 10 mg in patients with homozygous sitosterolemia: a 2-year, open-label extension study. Int J Clin Pract. 2008 Oct;62(10):1499-510. doi: 10.1111/j.1742-1241.2008.01841.x. PMID 18822021